CLINICAL TRIAL: NCT04584918
Title: An Open Label Study to Assess the Effect of Euryco-10® Oral Dietary Supplement on Total Testosterone, Sex Drive and Energy Level in Senior Men
Brief Title: An Open Label Study to Assess the Effect of Euryco-10® Oral Dietary Supplement in Senior Men
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Innovus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INNV-BHT1000-001
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Healthy Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the effect and support the tolerance of orally ingested formulation containing Eurycoma longifolia dietary supplement (Euryco-10) on a cohort of senior men.

DETAILED DESCRIPTION:
This is a single-center, single arm, open label study in senior men. This study will investigate the effect and tolerance of oral ingestion of Euryco-10. Subjects meeting all inclusion and none of the exclusion criteria will be enrolled and provided with study dietary supplement. Subjects will be instructed to take 2 capsules per day for 35 days. Administration and any adverse events will be recorded in the subject diary. At each clinic visit (Day 0, Day 21 and Day 35) the Subject will complete the AMS Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Male ≥ 55 years of age

Exclusion Criteria:

Severe lower urinary tract symptoms.

Current use of any herbal and/or nutritional supplements that can interfere with testosterone.

A history of cancer except melanoma skin cancer.

Currently receiving treatment with cancer chemotherapy or antiandrogens.

Chronic use of systemic glucocorticoids (use within >14 days up to the 3months prior to screening); use of non-testosterone anabolic steroids within12 months prior to screening.

History of frequent opioid use >1 time/week during any week within 30 days prior to screening.

Have a history of known angina.

Have a history of severe liver disease or clinical evidence of hepatic impairment at screening.

Untreated severe obstructive sleep apnea.

Allergies to any of the ingredients in Euryco-10® or BioPerine.

Any condition which would interfere with the subject's ability to provide informed consent, to comply with study instructions, or which might confound the interpretation of the study results

Min Age: 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum total testosterone concentration compared to baseline | Day 0, Day 21 and Day 35

SECONDARY OUTCOMES:
Change in Q 9 of the AMS Questionnaire | Day 0, Day 21 and Day 35
Change in Q17 of the AMS Questionnaire | Day 0, Day 21 and Day 35

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided